CLINICAL TRIAL: NCT00831337
Title: The Study of Probiotics in Liver Cirrhosis Patients With Portal Hypertension.
Brief Title: Evaluation of Probiotics in the Treatment of Portal Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Wojciech Marlicz, MD PhD, Pomeranian Medical University Szczecin
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PAM 12/06/PB
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Liver Cirrhosis; Portal Hypertension; Encephalopathy
Keywords: VSL3; Probiotics; Gut microbiota; Cytokines; Portal hypertension; Chemokines; Liver cirrhosis
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal; Brain Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Liver cirrhosis compensated (Experimental): VSL3 supplemented twice daily for 28 days
  Interventions: Dietary Supplement: VSL3
- Liver cirrhosis decompensated (Experimental): VSL3 supplemented twice daily for 28 days
  Interventions: Dietary Supplement: VSL3
- Control group (Experimental): VSL3 supplemented twice daily for 28 days
  Interventions: Dietary Supplement: VSL3

INTERVENTIONS:
Dietary Supplement: VSL3 — 2 times daily 450 billion live bacteria (in each saschet)

SUMMARY:
This study is to evaluate the role of probiotics in the treatment of portal hypertension. In particular the role of probiotics on gut microbiota in liver cirrhosis patients will be studied and compared with cytokines and other substances implicated in the pathogenesis of portal hypertension. The hypothesis whether probiotics may change the prognosis of patients with portal hypertension will be studied. The hypothesis whether probiotics may halt the pathologic cascade of events leading to various complications (e.g. hepato-renal syndrome, spontaneous bacterial peritonitis, bleeding varices) will be reviewed.

DETAILED DESCRIPTION:
Studied probiotics: VSL3

ELIGIBILITY:
Inclusion Criteria:

* Confirmed liver cirrhosis (liver biopsy or typical imaging studies)
* Confirmed portal hypertension
* 18 years and older
* compliant patients

Exclusion Criteria:

* Antibiotic treatment in last 3 months
* Lactulose treatment in last 3 months
* Patients taking NSAIDS in lat 3 months
* Steroid treatment in last 3 months
* Ongoing and active infection
* Pregnant woman
* Cancer diagnosis
* decompensated diabetes mellitus
* active or past treatment with recombinant cytokines (e.g. anty TNF, interferon etc)
* medication altering function of CNS, suffering from neurological or ophthalmological conditions
* initiating the therapy with beta blockers within the prior 12 weeks
* mental disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-04; Primary Completion 2010-11 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Laboratory data | 28 days

SECONDARY OUTCOMES:
Clinical and laboratory data | 1 months

CONTACTS AND LOCATIONS:
Overall Officials: Wojciech M Marlicz, M.D., Ph.D., Principal Investigator — Pomeranian Medical University Szczecin
Locations (1):
- Department of Gastroenterology, Pomeranian Medical University, Szczecin, Poland